CLINICAL TRIAL: NCT01134159
Title: Registry Experience at the WAshington Hospital CenteR, DeS - Taxus Liberte vs Xience V
Brief Title: Registry Experience at the Washington Hospital Center, Des - Taxus Liberte Versus Xience V
Acronym: REWARDS TLX
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Ron Waksman, M.D., Cardiovascular Research Institute/ Medstar Health Research Institute
Other Study IDs: REWARDS TLX
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Xience V: Those who have only received a Xience V stent
- Taxus Liberte: Those who have received only a Taxus Liberte stent

SUMMARY:
Multicenter, retrospective registry to collect 9-12 month follow-up data to evaluate major adverse cardiac events in patients whom have undergone percutaneous coronary intervention and received either Taxus Liberte or Xience V.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older, both genders
* Underwent PCI with Taxus Liberte (alone) or Xience (alone)

Exclusion Criteria:

* Underwent PCI with a non-Taxus Liberte or Xience V DES during the same procedure
* Received both Taxus-Liberte and Xience-V during the same index procedure
* Patients not taking, or unable to take, dual antiplatelet therapy (aspirin plus clopidogrel or prasugrel).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients male or female, 18 years or older whom have undergone PCI with either Taxus Liberte or Xience V
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events, | 1 year
  A composite of all-cause death, Q-wave myocardial infarction, and target vessel revascularization

SECONDARY OUTCOMES:
Stent thrombosis | 1 year
Target vessel revascularization | 1 year
Cardiac death | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (10):
- United States (10):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Iowa Heart Center, West Des Moines, Iowa
  - Maine Medical Center, Portland, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Grand Strand Regional Medical Center, Myrtle Beach, South Carolina
  - Heart Clinics Northwest, Spokane, Washington

REFERENCES:
- [Derived] Waksman R, Ghali M, Goodroe R, Ryan T, Turco M, Ring M, McGarry T, Dobies D, Shammas N, Steinberg DH, Swymelar S, Kaneshige K, Torguson R. Percutaneous coronary intervention with second-generation paclitaxel-eluting stents versus everolimus-eluting stents in United States contemporary practice (REWARDS TLX Trial). Am J Cardiol. 2012 Oct 15;110(8):1119-24. doi: 10.1016/j.amjcard.2012.05.050. Epub 2012 Jul 3. PMID 22762711